CLINICAL TRIAL: NCT06031883
Title: Efficacy of Adding Low Dose Ketamine or Fentanyl to Propofol-dexmedetomidine as Total Intravenous Anesthesia for Patients Undergoing Craniotomy
Brief Title: Efficacy of Adding Low Dose Ketamine or Fentanyl to Propofol-dexmedetomidine as Total Intravenous Anesthesia
Acronym: TIVA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minia University (Other)
Collaborators: Minia University Hospital (Other)
Responsible Party: Principal Investigator, Eron Ashraf Faried, Eron Ashraf Faried, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 685-2023
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-02

CONDITIONS: Patients Undergoing Elective Craniotomy
MeSH Terms: interventions — Ketamine; Fentanyl

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 1 (Experimental): Ketamine group recieve induction and maintenance doses of ketamine by target controlled infusion in addition of propofol-dexmedetomidine as total intravenous anesthesia for patients undergoing craniotomy
  Interventions: Drug: Ketamine
- 2 (Experimental): Fentanyl group recieve induction and maintenance doses of fentanyl by target controlled infusion in addition of propofol-dexmedetomidine as total intravenous anesthesia for patients undergoing craniotomy
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Total intravenous anesthesia in craniotomy
  Other Names: Fentanyl

SUMMARY:
Efficacy of adding low dose ketamine or fentanyl to propofol-dexmedetomidine as total intravenous anesthesia for patients undergoing craniotomy in supra tentorial brain tumor

DETAILED DESCRIPTION:
Efficacy of adding low dose ketamine or fentanyl to propofol-dexmedetomidine as total intravenous anesthesia for patients undergoing craniotomy in supra tentorial brain tumor surgery on brain relaxation score, hemodynamics, surgeon satisfaction score , total requirement of intra operative propofol and post operative analgesia

ELIGIBILITY:
Inclusion Criteria:

- Patients aged 18-70 years old ASA I - III with GCS 14-15 and BMI<35 scheduled for elective craniotomy for resection of supratentorial masses

Exclusion Criteria:

* Patients will be excluded if they will refuse to give a written consent. Also patients with GCS < 14 or having endocrine or blood diseases or sever cardiac disease or sever liver disease or renal failure and patients with uncontrolled hypertension or uncontrolled diabetes mellitus and patients have allergy to any of the study drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of brain relaxation score | Intraoperative
  1:perfectly relaxed , 2:satisfactory relaxed , 3:firm brain and 4:bulging brain

CONTACTS AND LOCATIONS:
Locations (1):
- Eron, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No